CLINICAL TRIAL: NCT03293563
Title: UroCCR Database: French Research Network for Kidney Cancer (National Multidisciplinary Clinical and Biological Database on Kidney Cancer)
Brief Title: UroCCR Database: French Research Network for Kidney Cancer -UroCCR
Acronym: UroCCR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2011/38
Record Dates: First submitted 2016-07-12; First posted 2017-09-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Kidney Cancer
Keywords: Kidney cancer; Surgical approaches; Medical treatment; Multicentric and multidisciplinary network
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Adult patients with kidney cancer
  Interventions: Procedure: Radical nephrectomy versus partial nephrectomy (according surgeon judgement)

INTERVENTIONS:
Procedure: Radical nephrectomy versus partial nephrectomy (according surgeon judgement)

SUMMARY:
Kidney cancer management has become increasingly complex with the diversification of treatment options and the integration of multidisciplinary care. To meet these challenges, the UroCCR network was established in France as a national registry and research platform dedicated to renal cancer. Funded by the French National Cancer Institute (INCa), UroCCR prospectively collects comprehensive real-world data on patient care and disease evolution, while systematically linking these records with annotated biological samples (plasma, urine, and both healthy and tumour tissues). For each case, more than one thousand variables may be recorded, covering clinical, imaging, and patient-reported information.

More than a registry, UroCCR is a collaborative network of clinical and research professionals using a shared, evolving tool that supports rapid implementation of studies and fosters active knowledge generation. Unlike retrospective registries or sample-centred biobanks, UroCCR offers prospective, patient-focused inclusion and a wide scope of investigation-from translational and technological research to clinical evaluation and social sciences. It also supports multiple ancillary studies, including retrospective analyses and prospective clinical or observational trials, and operates under a structured governance system with recognised national and international labels.

By combining a rigorously structured, multicentre dataset with linkage to the French national health data system (SNDS), the platform uniquely unites detailed clinical annotation with population-wide coverage, creating a high-value environment for advancing kidney cancer research and care.

DETAILED DESCRIPTION:
The UroCCR project is a national kidney cancer registry and research network designed to address the specific challenges of renal cell carcinoma (RCC) management. While general cancer registries such as FRANCIM provide valuable surveillance data, most large-scale registries lack the depth of clinical, biological, and longitudinal follow-up information necessary to advance research and enable comprehensive analyses of kidney cancer outcomes. UroCCR was created in 2011 to meet this need.

With over 21,000 cases collected from 58 centres across France, UroCCR is now one of the largest national databases dedicated to kidney cancer worldwide. The registry captures detailed clinical parameters, treatments and outcomes, complemented by patient-reported measures and socioeconomic data. Because management practices within UroCCR follow the recommendations of the French Association of Urology (AFU), the dataset closely reflects real-world practice and provides a reliable basis for comparison with national and European guidelines. Moreover, patient data can be reused across numerous studies, allowing researchers to explore multiple scientific questions without requiring new enrolments for each project.

A distinctive strength of UroCCR is its integration of multiple research dimensions. Beyond clinical outcomes, it evaluates quality of life and the social and economic impact of kidney cancer. The registry is linked to annotated biobanking and national medico-administrative datasets, enabling translational studies and health services research. Additionally, UroCCR supports multiple ancillary studies, both retrospective analyses based on real-world data and prospective studies including randomised clinical trials or observational cohorts.

The project benefits from robust governance structures, ensuring standardised procedures, data quality, and ethical oversight. It has also received various national and international labels, recognising its methodological rigour and excellence in research infrastructure.

Digital innovations developed within the network, such as UroConnect® for perioperative monitoring and UroPredict machine learning models for recurrence and survival prediction, highlight its commitment to advancing care through new technologies.

At the national level, projects such as CARARE are developing personalised treatment strategies, including a molecular tumour board for non-clear cell RCC. Internationally, UroCCR is strengthening collaboration through partnerships with the European Association of Urology and the European Robotic Urology Section, contributing to harmonised data collection and large-scale multicentre research.

Ultimately, UroCCR functions as a dynamic research platform that unites clinicians, researchers, and patients around a shared infrastructure. By combining detailed clinical data with translational research, digital health tools, structured governance, recognised labels, and international partnerships, it aims to generate increasingly precise insights into RCC and to support the development of more effective, personalised treatment strategies in France and worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with kidney cancer
* Patient with no opposition to collection of its data for the study

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Kidney cancer
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2011-12; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the rates of complications between radical nephrectomy and partial nephrectomy | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Operative time, ,
Comparison of the rates of complications between radical nephrectomy and partial nephrectomy | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Blood loss
Comparison of the rates of complications between radical nephrectomy and partial nephrectomy | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Clinical scores

SECONDARY OUTCOMES:
Dosage of creatininemia to assess the renal function after surgery | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Dosage of creatininemia
Dosage of MDRD GFR to assess the renal function after surgery | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Dosage of MDRD GFR
Comparison of the rates of mortality between radical nephrectomy and partial nephrectomy | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Medical or surgical complication rates with Clavien's grading
Comparison of the rates of mortality between radical nephrectomy and partial nephrectomy | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Medical or surgical complication rates with urinary fistula rate
Comparison of the rates of mortality between radical nephrectomy and partial nephrectomy | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Medical or surgical complication rates with necessity for nephrectomy or re-exploration
Safety and efficacy of medical treatment on kidney tumor size evolution | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Imaging data: tumor size evolution
Safety and efficacy of medical treatment on biological parameters | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Biological parameters
Progression of the tumor | At Month 3, Month 6, Month12, and then every year for 5 years and every 2 years for 10 years
  Imaging data: tumor location

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe BERNHARD, PHU, Principal Investigator — University Hospital, Bordeaux
Locations (58):
- Hopital Universitaire de Bruxelles, Brussels, Belgium
- France (55):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - Clinique TIVOLI-DUCOS, Bordeaux
  - Polyclinique Médipôle Saint-Roch_Cabestany, Cabestany
  - CHU Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Ch Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor - APHP, Créteil
  - CHU de Dijon et CLCC Dijon, Dijon
  - CH du Sud Seine et Marne, Fontainebleau
  - Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - CHU Grenoble, La Tronche
  - Pôle Santé Sud, Le Mans
  - CH Libourne, Libourne
  - CHRU Lille - Centre Oscar Lambret, Lille
  - Hôpital privé La Louvière, Lille
  - CHU Limoges, Limoges
  - HCL Lyon, Lyon
  - APH Marseille, Marseille
  - Institut Paoli-Calmette, Marseille
  - Centre Hospitalier d' Annecy Genevois, Metz
  - CH Mont de Marsan, Mont-de-Marsan
  - Clinique du Pont de Chaume, Montauban
  - CHRU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - Clinique Saint George, Nice
  - CHU de Nîmes, Nîmes
  - CHU d'Orléans, Orléans
  - CHU Kremlin Bicêtre - APHP, Paris
  - CH St Joseph, Paris
  - Hôpital Européen Georges Pompidou - APHP, Paris
  - CHU Tenon - APHP, Paris
  - Hôpital Bichat -APHP, Paris
  - Hôpital Cochin Port-Royal - APHP, Paris
  - Hôpital Pitié Salpétrière - APHP, Paris
  - Institut Mutualiste Montsouris, Paris
  - Polyclinique Francheville, Périgueux
  - Hôpital privé des Côtes d'Armor, Plérin
  - CHU Poitiers, Poitiers
  - Hôpital privé Claude Galien, Quincy-sous-Sénart
  - Clinique La Croix Du Sud, Quint-Fonsegrives
  - CHU Reims, Reims
  - CHU Rennes - Centre Eugène Marquis, Rennes
  - CHU Rouen, Rouen
  - CHU St-Etienne, Saint-Etienne
  - Clinique Santé Atlantique de Nantes, Saint-Herblain
  - Clinique Urologique Nantes Atlantis, Saint-Herblain
  - Clinique Belledonne, Saint-Martin-d'Hères
  - CHU Strasbourg, Strasbourg
  - ICANS, Strasbourg
  - CHU Toulouse - Centre Claudius Régaud, Toulouse
  - Clinique Pasteur, Toulouse
  - CHRU Tours, Tours
  - Institut de Cancérologie lorraine, Vandœuvre-lès-Nancy
- Centre Hospitalier de Kourou, Kourou, French Guiana
- CHU Bellepierre, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Binzaqr S, Kryza D, Giraudet AL, Bernhard JC, Gross-Goupil M, Yacoub M, Margue G, Hindie E, Morgat C. Prostate-specific membrane antigen (PSMA) expression in primary and metastatic renal cell cancer (UroCCR-65 study). EJNMMI Res. 2025 Apr 9;15(1):38. doi: 10.1186/s13550-025-01232-8. PMID 40205264
- [Derived] Ingels A, Bensalah K, Beauval JB, Paparel P, Roupret M, Lang H, Nouhaud FX, Henon F, Bruyere F, Audenet F, Lebacle C, Baumert H, Long JA, Tambwe R, Charles T, Xylinas E, Waeckel T, Michiels C, Asselineau J, Benard A, Margue G, Boissier R, Bigot P, Bernhard JC; Comite Cancer de l'Association Francaise d'Urologie (CCAFU). Comparison of open and robotic-assisted partial nephrectomy approaches using multicentric data (UroCCR-47 study). Sci Rep. 2022 Nov 8;12(1):18981. doi: 10.1038/s41598-022-22912-8. PMID 36347900
- [Derived] Morrone A, Bentellis I, Bernhard JC, Bensalah K, Champy C, Bruyere F, Doumerc N, Olivier J, Audenet F, Parier B, Brenier M, Long JA, Nouhaud FX, Branger N, Lang H, Charles T, Xylinas E, Waeckel T, Gomez F, Boissier R, Rouget B, Shaikh A, Chevallier D, Ambrosetti D, Durand M. Positive surgical margin's impact on short-term oncological prognosis after robot-assisted partial nephrectomy (MARGINS study: UroCCR no 96). Sci Rep. 2022 Oct 31;12(1):18342. doi: 10.1038/s41598-022-23146-4. PMID 36316438
- [Derived] Brehier G, Bouvier A, Besnier L, Willoteaux S, Nedelcu C, Culty T, Aube C, Bigot P. Renal function after partial nephrectomy following intra-arterial embolization of renal tumors. Sci Rep. 2020 Dec 7;10(1):21352. doi: 10.1038/s41598-020-78461-5. PMID 33288819
- See also: Program I.Care Bordeaux — https://icare-bordeaux.fr/programme-i-care/
- See also: UroPredict Algorithm — https://uropredict.sophiagenetics.com/?model=uropredict1